CLINICAL TRIAL: NCT06889701
Title: A Phase 1/2 Study to Evaluate the Safety, PK and Efficacy of TNP-2092 Administered Via IA Injection in Participants With Early or Acute Hematogenous PJI Requiring or Not Requiring DAIR After TKA, or Requiring Long-term Antibiotic Therapy
Brief Title: A Phase 1/2 Study to Evaluate the Safety, PK and Efficacy of TNP-2092 Administered Via IA Injection in PJI Participants
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TenNor Therapeutics Inc. (Industry)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNP-2092-IA-01
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Periprosthetic Joint Infection (PJI)
MeSH Terms: interventions — TNP-2092; Injections; Vancomycin; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Three eligible participants will be enrolled as sentinel group. After all sentinel participants are tolerable safety at EA assessment and complete the PK study, an additional 20 participants will be enrolled and randomize in 1:1 ratio to the experimental group and the control group.
  Ten subjects requiring long-term suppressive antibiotic therapy for PJI (including PJI occurring after various joint replacement surgeries) will be enrolled in the expansion group and could be enrolled in parallel with the sentinel group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sentinel group (Experimental): In the sentinel group, participants will receive TNP-2092 50 mg IA+vancomycin IV+oral antibiotics.
  Interventions: Drug: TNP-2092 for injection; Drug: Vancomycin Hydrochloride for Injection (IV); Drug: Oral antibiotics
- Experimental group (Experimental): In the experimental group, participants will receive TNP-2092 50 mg IA + vancomycin IV + oral antibiotics.
  Interventions: Drug: TNP-2092 for injection; Drug: Vancomycin Hydrochloride for Injection (IV); Drug: Oral antibiotics
- Control group (Active Comparator): In the control group, participants will receive vancomycin IA + vancomycin IV + oral antibiotics.
  Interventions: Drug: Vancomycin Hydrochloride for Injection (IA); Drug: Vancomycin Hydrochloride for Injection (IV); Drug: Oral antibiotics
- Expansion group (Experimental): In the expansion group, participants will receive TNP-2092 50 mg IA based on the background treatment.
  Interventions: Drug: TNP-2092 for injection; Drug: Background Treatment

INTERVENTIONS:
Drug: TNP-2092 for injection — TNP-2092 for injection, 100 mg/vial, Intra-articular administration (IA), 10ml (50 mg) once daily for 14 days. TNP-2092 dose volume, dose, frequency, and duration can be adjusted according to the sentinel group synovial fluid TNP-2092 concentration, PK characteristics, and safety results at the EA visit.
  Other Names: rifaquizinone for injection
  Arms: Expansion group; Experimental group; Sentinel group
Drug: Vancomycin Hydrochloride for Injection (IA) — Vancomycin Hydrochloride for Injection, 0.5 g/vial, Intra-articular administration, 10 mL (0.5 g) once daily for 14 days.
  Arms: Control group
Drug: Vancomycin Hydrochloride for Injection (IV) — Vancomycin Hydrochloride for Injection, 0.5 g/vial, Intravenous infusion, 250 mL (1 g) q12h ± 1h per day, for 14 days.
  Arms: Control group; Experimental group; Sentinel group
Drug: Oral antibiotics — Rifampicin capsules: 0.15 g/capsule. 0.45 g (3 capsules) orally once daily within 1 h before breakfast for 8 weeks (56 days).
  Levofloxacin Tablets: 0.5 g/tablet. 0.5 g (1 tablet) orally once daily within 1 hour before breakfast for 8 weeks (56 days).
  If susceptibility testing results show resistance to rifampicin and/or levofloxacin, or intolerance by the patient 's participant, treatment with oral minocycline hydrochloride capsules will be substituted as follows:Minocycline hydrochloride capsules: 100 mg/capsule. Administered orally q12h ± 1h daily, doubling the first dose, 200 mg (2 capsules) orally, then 100 mg (1 capsule) each time for 8 weeks (56 days).
  The total duration of oral treatment during the oral administration period was 8 weeks (56 days) regardless of whether oral medication will be changed (eg, intolerance).
  Arms: Control group; Experimental group; Sentinel group
Drug: Background Treatment — Background treatment will be determined by the investigator.
  Arms: Expansion group

SUMMARY:
This is a Phase 1/2, randomized, controlled, open-label, proof-of-concept study to evaluate the safety and tolerability, local and systemic PK profiles of TNP-2092 administered via IA injection on the basis of vancomycin IV and oral antibiotics therapy in participants with early (within 1 month of TKA) or acute hematogenous (within 3 weeks of infectious symptoms) PJI requiring or not requiring DAIR therapy after TKA, or requiring long-term antibiotic suppression therapy for PJI (including PJI occurring after various joint replacements and revision surgeries).

DETAILED DESCRIPTION:
The study population is participants with confirmed or suspected Gram-positive bacteria causing early (ie, within 1 month of TKA) or acute hematogenous (within 3 weeks of infection symptoms) PJI requiring or not requiring DAIR therapy following TKA, or requiring long-term antibiotic suppression therapy for PJI (including PJI occurring after various joint replacement and revision surgeries). Participants will undergo screening assessments within 7 days prior to study start.

ELIGIBILITY:
Inclusion Criteria:

* Early (within 1 month of TKA) or acute hematogenous (within 3 weeks of infectious symptoms) PJI requires or does not require DAIR therapy after TKA, or results of treatment for PJI (including PJI occurring after various joint replacements and revision surgeries) did not meet the clinical cure criteria and requiring long-term antibiotic suppression therapy as judged by investigators before enrollment.
* Suspected or confirmed PJI was caused by a Gram-positive bacterial infection, including methicillin-resistant and ciprofloxacin-resistant Staphylococcus aureus and Staphylococcus epidermidis, as judged by the investigator.
* Agree to be hospitalized for 2 weeks with local intra-articular injection.
* 18 years of age or older (of either sex) at the time of signing the informed consent form (ICF).
* The implanted prosthetic joint was well fixed.
* No sinus tract that communicates with the prosthesis.
* Body mass index (BMI) ≥ 18 kg/m^2 and ≤ 34 kg/m^2.
* Agree to voluntarily use effective contraception from signing the ICF through 8 weeks after the last dose of investigational product (in case of premature withdrawal from the study) or through completion of the end-of-study visit. Male participants must refrain from donating sperm during this period.

Exclusion Criteria:

* History of hypersensitivity or intolerance to any of the following agents: vancomycin or TNP-2092.
* Definite PJI of Gram-negative infection, fungal infection, or Enterococcus infection, or Mycobacterium infection, or Gram-positive mixed Gram-negative and/or fungal infection.
* Definite systemic infection (sepsis).
* Expected survival less than 1 years.
* Female participant is pregnant, lactating, or has a positive screening/baseline pregnancy test.
* Surgical or medical conditions that, in the opinion of the investigator, could affect the participant's ability to participate in the study, or affect the administration of investigational product, or affect the interpretation of study results, including but not limited to active malignancy, metabolic disease, alcohol or drug abuse, or clinically significant laboratory abnormalities.
* Presence of serious liver, blood, or immune system disorders as evidenced by the following:

  1. Acute hepatitis of any cause within the past year.
  2. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels > 2 times the upper limit of normal (ULN).
  3. Presence of end-stage liver disease-related manifestations such as ascites or hepatic encephalopathy.
  4. Current or anticipated neutropenia (ie, neutrophil count < 0.5 x 10^9/L).
  5. Chemotherapy for cancer, radiation therapy, or potent noncorticosteroid immunosuppressants (eg, cyclosporine, azathioprine, tacrolimus, immunomodulatory monoclonal antibody therapy, etc) within the past 3 months or corticosteroids (≥ 40 mg prednisone/day) for more than 14 days within 30 days prior to randomization.
* Positive AIDS antibody screening.
* History or evidence of severe renal disease or creatinine clearance < 30 mL/min based on the Cockcroft-Gault formula.
* Treatment with an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Participants who, in the opinion of the investigator, were unable to comply with the protocol and study drug administration procedures or complete the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of TNP-2092 by Assessment of the Number of Adverse Events (AEs) | Day 1 to Day 187
  An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
TNP-2092 concentrations in synovial fluid | At 12, 24 hours after the first dose of TNP-2092, before dosing on Day 7, before the last dose, and at 12, 24, 48 hours after the last dose.
  Synovial fluid concentrations of TNP-2092 were measured by a specific and validated assay.
Maximum Observed Plasma Concentration (Cmax) of TNP-2092 after the first dose | Before administration (within 1 hour), 1, 4, 12, 24 hours after the first dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) after the first dose | Before administration (within 1 hour), 1, 4, 12, 24 hours after the first dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area under the curve from the time of dosing to the last measurable concentration (AUC 0-t) after the first dose | Before administration (within 1 hour), 1, 4, 12, 24 hours after the first dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area under the curve from the time of dosing to infinity (AUC 0-∞) after the first dose | Before administration (within 1 hour), 1, 4, 12, 24 hours after the first dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Elimination half-life (t 1/2) after the first dose | Before administration (within 1 hour), 1, 4, 12, 24 hours after the first dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Maximum observed concentration at steady state (Cmax, ss) after the last dose | Before administration (within 1 hour), 1, 4, 12, 24, 48 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time to maximum concentration at steady state (Tmax, ss) after the last dose | Before administration (within 1 hour), 1, 4, 12, 24, 48 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area under the curve from the time of dosing to the last measurable concentration at steady state (AUC 0-t, ss) after the last dose | Before administration (within 1 hour), 1, 4, 12, 24, 48 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area under the curve from the time of dosing to infinity at steady state (AUC 0-∞, ss) after the last dose | Before administration (within 1 hour), 1, 4, 12, 24, 48 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area under the curve over the dosing interval at steady state (AUC 0-tau, ss) | Before administration (within 1 hour), 1, 4, 12, 24 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Elimination half-life at steady state (t 1/2, ss) | Before administration (within 1 hour), 1, 4, 12, 24, 48 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Accumulation ratio (Rac) | Before administration (within 1 hour) of the first dose, 1, 4, 12, 24 hours after the first dose; Before administration (within 1 hour) of the last dose, 1, 4, 12, 24 hours after the last dose
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Early Assessment (EA) response rate | Day 14
  Participants with early or acute hematogenous PJI after TKA who met all the following criteria will be judged as responders:
  * At least 2 body temperature measurements within the last 24 hours separated by more than 6 hours were ≤ 37.6ºC.
  * Peripheral white blood cell (WBC) count returned to normal range (as determined by local laboratory reference range).
  * Synovial fluid WBC < 3000 cell/μL and polymorphonuclear leukocytes percentage (PMN%) < 80%.
  * Inflammatory manifestations (pain, erythema, edema, wound exudate) at the primary infection site resolved, with pain requiring resolution or tolerance.
  * Inflammatory markers (ie, C-reactive protein [CRP]) improved to 50% of normal or baseline values.
End of treatment (EOT) response rate | Day 71 to Day 77
  Participants who met all the following criteria were judged as responders:
  * Joint pain resolved or tolerated.
  * Joint function improvement.
  * Inflammatory markers (ie, CRP) returned to ≤ 10 mg/L.
Treatment failure rate | Within 6 months after the start of study treatment
  Those who meet any of the following criteria are treatment failures:
  * No response at EA assessment (only for participants with early or acute hematogenous PJI after TKA).
  * No response at EOT assessment.
  * Receiving systemic antibiotics for infected joints after the end of study treatment.
  * Additional surgical treatment of infected joints is required during the study.
  * Death due to primary joint infection.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT06889701/Prot_001.pdf